CLINICAL TRIAL: NCT05067322
Title: Therapeutic Gaming for the Treatment of Attention Deficit Hyperactivity Disorder
Acronym: THERAGAME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment at the site.
Sponsor: Spherix Incorporated (Industry)
Collaborators: BioSpherix (Industry)
Responsible Party: Principal Investigator, Robert A Lodder, PhD, Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: TVG001
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Test group and a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minecraft (Experimental): This group played the video game under development in Minecraft
  Interventions: Device: Minecraft
- Control (Placebo Comparator): This group played another game.
  Interventions: Device: Minecraft

INTERVENTIONS:
Device: Minecraft — A game played within the videogame Minecraft

SUMMARY:
Children with ADHD play a videogame to test symptom control

DETAILED DESCRIPTION:
Minecraft is an online video game containing a "virtual land where users can create their own worlds and experiences, using building blocks, resources discovered on the site and their own creativity" that requires its users to apply problem solving, planning, and organizational skills for creative building and exploration.1

It is being studied as an adjunctive treatment in combination with stimulant medications in children with attention deficit hyperactivity disorder (ADHD) to improve executive function and ADHD symptoms, as well as to allow for the use of lower doses of stimulant drugs. Although there is little research on the effect of Minecraft in humans, there is considerable research on the effects of other video games. Like pharmaceuticals, the effect seen seems to be often related to the amount and style of video games to which humans are exposed. First-person shooter games with violence have been associated with anxiety and fear (Strasburger et al. 2010). The negative outcomes of video play include obesity, aggressiveness, antisocial behavior, and addiction (Strasburger et al 2010).2 Video and computer games come in many different genres, some violent, some nonviolent, some with lots of action, some without any action, etc. Chess and checkers were among the earliest computer games and they still remain popular. Cognitive training interventions administered in a game format have been studied in children with ADHD. Taken together, the results of studies show that these cognitive training interventions are generally effective in improving the specific executive functions they target, as well as parent-reported ADHD symptoms. The majority of the interventions studied have targeted training of working memory, although some interventions have also targeted attention, response inhibition, and cognitive flexibility in the training. A recent meta-analysis found that interventions targeting multiple executive function domains had a stronger effect on parent-reported ADHD symptoms than studies targeting working memory alone (which showed minimal benefits), but it is possible that the greater benefits seen were due to a more intensive intervention schedule.3

The improvements in cognitive assessments and parent-rated ADHD symptoms have been shown to persist for up to 6 months after completion of training.4 However, it should be noted that the improvements in cognitive function could be due to practice effects arising from repetition of the cognitive tasks, rather than a true alteration in cognitive function.5 In contrast to the effects on "near-transfer" functions and parent-rated ADHD symptoms, evidence of "far-transfer" effects to untrained functions and non-clinical environments has been limited, and improvements in teacher-rated ADHD symptoms have not been observed. The latter observation is particularly important as teacher ratings of ADHD symptoms can be a more objective measure of efficacy than parent ratings, and the most significant limitations for a majority of the studies have been effective blinding procedures and an appropriate control condition. These results are further limited by overrepresentation of males subjects in study populations, the exclusion of patients with comorbidities in most of the studies, and small sample sizes (for review, see Rutledge, et al. (2012), Chacko, et al. (2013) , and Rivero, et al. (2015)).

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary diagnosis of ADHD in accordance with DSM-5. 2. On a current regimen of a stimulant type ADHD medication, such as Vyvanse. 3. Sex: males and females. 4. Age: between 10 and 15 years of age. 5. Stated willingness to comply with all study procedures and availability for the duration of the study, including adherence to medication and play regimen. 6. Are capable, as determined by the investigator, to perform the following:

  1. complete the study log.
  2. are able to comply with the required study visits. 7. Have given written informed assent along with parents/legal guardians to participate in this study in accordance to local regulations before any trial related activities (other than initial screening) are carried out. 8. Are Minecraft players and have access to a full version of PC/Mac (Java) Minecraft, Xbox Minecraft, or pocket Minecraft version (Android, Kindle) that supports play on Realms. 9. Subjects' parents and subjects both currently have Google accounts and electronic devices to access Google accounts online. 10.Must have an NICHQ Vanderbilt Assessment scored by parents and teacher(s) within the last month, or get an assessment scored by parents and teacher(s) within one week of enrollment and before beginning to play the video game if the subject is in the video game arm). 11.At least one parent and the subject must be proficient in spoken and written English.

Exclusion Criteria:

- 1. Current or past history of substance abuse. 2. Patients who for whatever reason are deemed by the investigator inadequate for participation in this trial (e.g., patients with incapacitating mental illness).

3. Have previously completed or withdrawn from this study after having signed the informed consent/assent document. 4. Lack of proficiency in spoken and written English

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Score on NICHQ Vanderbilt assessment | One month
  Score on NICHQ Vanderbilt assessment